CLINICAL TRIAL: NCT02747823
Title: A Randomized, Double-blind, Single-dose, 3-way, Parallel Group, Comparator-controlled, Adaptive Design, Pharmacokinetic, Safety, and Tolerability Study in Healthy Male Volunteers to Evaluate Bioequivalence of CBT124 to Avastin® (EU and US)
Brief Title: PK Bioequivalence Single-dose Safety Tolerability Study in Healthy Male Volunteers to Compare CBT124 & Avastin(EU&US)
Acronym: CBT124NHV001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cipla BioTec Pvt. Ltd. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: CBT124/NHV/001; ACTRN12616000428460 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CBT124 (Experimental): CBT124, single dose of 1 mg/kg, IV infusion
  Interventions: Biological: CBT124
- EU Sourced Avastin® (Active Comparator): EU Sourced Avastin®, single dose of 1 mg/kg, IV infusion
  Interventions: Biological: EU Sourced Avastin®
- US Sourced Avastin® (Active Comparator): US Sourced Avastin®, single dose of 1 mg/kg, IV infusion
  Interventions: Biological: US Sourced Avastin®

INTERVENTIONS:
Biological: CBT124 — 1 mg/kg IV infusion
  Arms: CBT124
Biological: EU Sourced Avastin® — 1 mg/kg IV infusion
  Arms: EU Sourced Avastin®
Biological: US Sourced Avastin® — 1 mg/kg IV infusion
  Arms: US Sourced Avastin®

SUMMARY:
This study aims to investigate the bioequivalence of new formulation of bevacizumab called CBT124 and safety when compared to two already marketed formulations, one approved in US and other in EU of Avastin(Registered Trademark). Adult healthy male aged 18 to 50 years (both inclusive) can participate in this trial.

Participants will be randomised (allocated by chance) to either a test formulation or one of the two marketed formulations of bevacizumab. Drugs will be administered intravenously once only. The study will compare the safety, tolerability, pharmacokinetics (PK) (the levels of drug in the blood), pharmacodynamics (PD) (what the drug does to the body) and immunogenicity (body's immune response) of the 3 drugs. In order to measure this, blood samples will be collected at various points after treatment has been given.

DETAILED DESCRIPTION:
Cipla BioTec, a pharmaceutical company (company developing drugs), is developing its own formulation of bevacizumab called CBT124 which is similar to Avastin(Registered Trademark). The formulation is, intended for intravenous (into a vein) administration for the treatment of certain cancers. CBT124 is also a type of monoclonal antibody with a proposed biological activity similar to bevacizumab. Research on CBT124 indicates that it should act the same as Avastin(Registered Trademark) in the body. It is expected that CBT124 will provide all the clinical advantages of the marketed drug Avastin(Registered Trademark). The main purpose of this study is to test that whether CBT124 behaves the same in the human body as Avastin(Registered Trademark) i.e. produce the same amount/concentration of drug in the blood as the EU and USA marketed drug, Avastin(Registered Trademark). This is called a 'biosimilar' study. The study will compare the safety, tolerability, pharmacokinetics (PK) (the levels of drug in the blood), pharmacodynamics (PD) (what the drug does to the body) and immunogenicity (body's immune (body's defense system) response) of the 3 drugs when given intravenously (into a vein) to healthy male participants: new drug called CBT124, marketed drug Avastin(Registered Trademark) approved in United States (US), marketed drug Avastin(Registered Trademark) approved in European Union (EU). The results will be compared to see if these drugs behave the same and are therefore equivalent. In order to measure this, blood samples will be collected after treatment has been given and the amount of drug in the blood measured at specific times. In addition, the study will also compare and analyse the effect the drug has on your immune system from blood samples. Safety and tolerability of both drugs will also be monitored and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy male subjects between 18.0 and 30.0 kg/m2 body mass index (inclusive) and body weight ≥ 60kg and ≤ 100 kg (inclusive)
2. Subjects who are healthy as determined by pre-study medical history, physical examination, vital signs and 12-lead ECG at screening and admission
3. Subjects whose clinical laboratory test results are normal, or where outside the reference range is judged as not clinically relevant by the Investigator
4. Have systolic blood pressure ≤ 140 and ≥ 90 mmHg
5. Have physical examination results without clinically relevant findings at screening and admission
6. Have 12-lead ECG results without clinically relevant findings at screening and admission
7. Subjects who are non-smokers and have not regularly used tobacco or nicotine containing products
8. Males must be willing to use a medically acceptable method of contraception from the time of the administration of investigational product (IP), throughout the study
9. Must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures
10. Must be able to provide informed consent which must be obtained prior to any study related procedures

Exclusion Criteria:

1. Have a history of hypersensitivity or allergic reactions
2. Have a history of or presence of current clinically significant gastrointestinal disorder
3. Have a history of and/or current cardiac disease
4. Have a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus, or human immunodeficiency virus (HIV) I and II at screening
5. Have a history of cancer
6. Have an illness within 30 days prior to screening, or prior to dosing, that is classed as clinically significant by the Investigator
7. Prior exposure to any investigational monoclonal antibody
8. Any clinically significant infection, in the opinion of the Investigator, ongoing at screening or admission to the clinical unit
9. Have had major surgery
10. Have received live vaccine(s)
11. Have an intake of alcoholic beverages
12. Have reasonable evidence of drug abuse as indicated by a positive urinary drug test at screening or admission
13. Have taken medication
14. Have donated > 100 mL blood within 4 weeks prior to the administration of the study drug
15. Have participated in another clinical study of an investigational drug
16. Subjects who, in the opinion of the Investigator, are not likely to complete the study for whatever reason
17. Impaired liver function as determined by: Serum alanine aminotransferase and/or aspartate aminotransferase > 1.5 x upper limit of normal (ULN) at screening or admission. Subjects with values between ULN and 1.5 x ULN may be included in the study if considered not clinically significant by the Investigator

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma | from 0 (baseline) up to 95 days extrapolated infinity (AUC(0 - ∞))

SECONDARY OUTCOMES:
Area under the concentration-time curve | from time 0 to the last quantifiable data point (AUC0-t)
Maximum observed plasma concentration (Cmax) | from time 0 to the last quantifiable data point (AUC0-t)
Time to maximum observed concentration (tmax) | from time 0 to the last quantifiable data point (AUC0-t)
Terminal half-life (t½) | from time 0 to the last quantifiable data point (AUC0-t)
Terminal rate constant (λz) | from time 0 to the last quantifiable data point (AUC0-t)
Systemic clearance (CL) | from time 0 to the last quantifiable data point (AUC0-t)
Volume of distribution at steady state (Vss) | from time 0 to the last quantifiable data point (AUC0-t)
Immunogenicity will be assessed by the incidence of anti-bevacizumab antibodies (ADA), including neutralizing antibodies (nAb) | Day 1 through last volunteer last visit
Safety and tolerability will be assessed by clinical laboratory tests, vital signs, 12-lead ECGs, physical examinations, assessment of adverse events (AE), injection site reactions and concomitant medications | Day 1 through last volunteer last visit

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schwabe, MD(GenSur), Principal Investigator — Auckland Clinical studies; Sepehr Shakib, MBBS,FRACP, Principal Investigator — c/o CMAX - a division of IDT Australia Ltd.
Locations (1):
- Auckland Clinical Studies Ltd., 3 Ferncroft Street, Grafton, Auckland, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
As sponsors, we would be protecting the confidentiality of the subjects and would be unaware of the IPD ourselves.